CLINICAL TRIAL: NCT02201004
Title: A Randomized, Double Blind Placebo Controlled 2-Arm Parallel Group, Multicenter Study With A 16-Week Treatment Assessing The Efficacy And Safety, And 52-Week Long Term Safety Including 36-Week Open Label Extension Of Tofogliflozin With Insulin Treatment In Type 2 Diabetes Mellitus
Brief Title: TOFO Insulin Combination Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOFOGL07061; U1111-1159-5316 (UTN)
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-((4-ethylphenyl)methyl)-3',4',5',6'-tetrahydro-6'-(hydroxymethyl)spiro(isobenzofuran-1(3H),2'-(2H)pyran)-3',4',5'-triol; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tofogliflozin (Experimental): Tofogliflozin administered once daily for 52 weeks. Insulin administered as base treatment.
  Interventions: Drug: TOFOGLIFLOZIN CSG452; Drug: insulin
- placebo (Placebo Comparator): Placebo administered once daily for 16 weeks. After 16-weeks, Tofogliflozin administered once daily for 36 weeks. Insulin administered as base treatment.
  Interventions: Drug: TOFOGLIFLOZIN CSG452; Drug: insulin; Drug: placebo

INTERVENTIONS:
Drug: TOFOGLIFLOZIN CSG452 — Pharmaceutical form:tablet Route of administration: oral
  Other Names: Apleway; Deberza
Drug: insulin — Pharmaceutical form:solution Route of administration: subcutaneous
Drug: placebo — Pharmaceutical form:tablet Route of administration: oral
  Arms: placebo

SUMMARY:
Primary Objectives:

To assess the effects of tofogliflozin on glycemic control in comparison to placebo as an add-on treatment to insulin treatment in terms of glycated hemoglobin (HbA1c) reduction over a period of 16 weeks in patients with type 2 diabetes mellitus.

To assess the safety of tofogliflozin in combination with insulin treatment throughout 52 weeks.

Secondary Objectives:

To assess the effects of tofogliflozin in comparison to placebo on:

* Body weight
* Fasting plasma glucose (FPG)
* Postprandial plasma glucose (PPG) To assess the long term safety and tolerability of tofogliflozin.

DETAILED DESCRIPTION:
The total study duration from screening for a patient can be approximately up to 1 year, including a screening period of 2 weeks, double-blinded placebo controlled treatment period of 16 weeks, an open-labeled extension period of 36 weeks, and a follow-up period of 3 days.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 20-75 years old with type 2 diabetes mellitus (T2DM).
* Hemoglobin A1c ≥7.5% - ≤10.5% and FPG ≤220 mg/dL.
* Basal bolus (BB), Bolus, Premix, Basal supported oral therapy (BOT) regimens used for more than 12 weeks before screening.
* Stable dose (-/+20%) of insulin and no change in the dose of oral hypoglycemic agents for more than 12 weeks before screening.
* Only Dipeptidyl peptidase-4 inhibitor is allowed for basal supported oral therapy (BOT) regimen.
* Body mass index (BMI) ≥18.5 kg/m^2 and <35.0 kg/m^2.
* No change of antihypertensive, anti-hypercholesterolemia and uric acid lowering drug 4 weeks before screening.

Exclusion criteria:

* Type 1 diabetes mellitus.
* Pregnancy or lactation.
* Severely uncontrolled glycemic situation.
* History of metabolic acidosis, including diabetic ketoacidosis, within 1 year prior to screening.
* History of myocardial infarction, stroke, or heart failure requiring hospitalization or drug or alcohol abuse within the previous 6 months.
* A measured serum creatinine level greater than 2.0 mg/dL for men and 1.5 mg/dL for women.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2.5 times the upper limit of the reference range at the central laboratory test facility.
* Has previously received treatment with the investigational product.
* Has received treatment with another investigational product or non-approved drug within 3 months before tests for provisional enrolment.
* Corticosteroid therapy for 14 or more days in total within 8 weeks before tests for provisional enrolment (excluding those used for localized effects, such as drugs for topical [skin] application, eye drops and sprays).
* Patients who are frequently experiencing orthostatic hypotension.
* Required a change in the dosing regimen for the following drugs within 4 weeks before tests for provisional enrolment:
* Lipid-lowering drug
* Antihypertensive drug
* Thyroid hormone preparation
* Uric acid lowering drug

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | 16 weeks after first intake of investigational product

SECONDARY OUTCOMES:
Change of Body Weight (BW) from baseline | 16 weeks after first intake of investigational product
Change of FPG from baseline | 16 weeks after first intake of investigational product
Change of PPG from baseline | 16 weeks after first intake of investigational product
Number of subjects with adverse events | Up to 52 weeks from the first intake of investigational medicinal product

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (30):
- Japan (30):
  - Investigational Site Number 392-028, Adachi-ku
  - Investigational Site Number 392-007, Atsugi-shi
  - Investigational Site Number 392-026, Chuoh-ku
  - Investigational Site Number 392-021, Fukuoka
  - Investigational Site Number 392-002, Ichihara-shi
  - Investigational Site Number 392-012, Iruma-shi
  - Investigational Site Number 392-003, Kawaguchi-shi
  - Investigational Site Number 392-014, Kitakyusyu-shi
  - Investigational Site Number 392-027, Kobe
  - Investigational Site Number 392-004, Koga-shi
  - Investigational Site Number 392-022, Kunitachi-shi
  - Investigational Site Number 392-019, Kurume-shi
  - Investigational Site Number 392-001, Kyoto
  - Investigational Site Number 392-024, Kyoto
  - Investigational Site Number 392-006, Matsudo-shi
  - Investigational Site Number 392-008, Mito
  - Investigational Site Number 392-030, Musashino-shi
  - Investigational Site Number 392-029, Okayama
  - Investigational Site Number 392-017, Ōtsu
  - Investigational Site Number 392-011, Sagamihara-shi
  - Investigational Site Number 392-020, Sakaishi
  - Investigational Site Number 392-010, Sapporo
  - Investigational Site Number 392-016, Sendai
  - Investigational Site Number 392-018, Shinjuku-ku
  - Investigational Site Number 392-005, Shizuoka
  - Investigational Site Number 392-031, Suita-shi
  - Investigational Site Number 392-015, Sumida-ku
  - Investigational Site Number 392-023, Sunto-gun
  - Investigational Site Number 392-013, Tokorozawa-shi
  - Investigational Site Number 392-025, Yokohama

REFERENCES:
- [Result] Terauchi Y, Tamura M, Senda M, Gunji R, Kaku K. Efficacy and safety of tofogliflozin in Japanese patients with type 2 diabetes mellitus with inadequate glycaemic control on insulin therapy (J-STEP/INS): Results of a 16-week randomized, double-blind, placebo-controlled multicentre trial. Diabetes Obes Metab. 2017 Oct;19(10):1397-1407. doi: 10.1111/dom.12957. Epub 2017 Jul 13. PMID 28371205